CLINICAL TRIAL: NCT00929032
Title: The Impact of Liver Transplantation on Reticuloendothelial Clearance Capacity
Brief Title: Liver Transplantation and Reticuloendothelial Clearance Capacity
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); European Society of Organ Transplantation (Unknown)
Responsible Party: The Queen´s Medical Research Institute, University of Edinburgh
Other Study IDs: NanospheresLiverEdinburgh09
Record Dates: First submitted 2009-06-24; First posted 2009-06-26 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-10

CONDITIONS: Hepatic Insufficiency; Liver Insufficiency
Keywords: Liver Transplantation; Immunosystem of the Liver; Marginal and Non-marginal grafts
MeSH Terms: conditions — Hepatic Insufficiency; Margins of Excision | interventions — technetium Tc 99m nanocolloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver transplant recipient: Liver transplant recipient
  Interventions: Radiation: Nanocoll®

INTERVENTIONS:
Radiation: Nanocoll® — To determine reticuloendothelial system (RES) phagocytosis activity and liver phagocytic function respectively we will measure plasma clearance of 99mTc labelled micro-aggregated human albumin without any imaging studies.

SUMMARY:
Study summary: "Liver transplantation and the reticuloendothelial clearance capacity."

The purpose of this study is to evaluate the effect of liver transplantation on the immune system.

This study will involve the taking of a number of observations but does not involve any treatment, which differs from normal care. Indications for transplantation are solely based on the best clinical practice, which is usually performed at the department.

The study measures liver function based on the clearance of different "marker" substances by the liver. These substances are given intravenously and their clearance will be measured from bloodstream.

All substances used in this study are registered in the United Kingdom for clinical applications and already used in clinical practice over years. They are safe and without any risk to harm individuals under study. Furthermore no side effects or any symptoms caused by the administration of these substances are expected.

Measurements of liver function are undertaken before transplantation, 1 and 7 days following the transplant. There is no restriction from any of the patient's prescribed medication. All blood samples will be removed from the cannula (drip) and will not require repeated injections. It is hoped that this research will lead to a greater understanding of the effects of liver transplantation on the immune system.

DETAILED DESCRIPTION:
Introduction

Liver cells called hepatocytes undertake the most important metabolic functions of the liver. The liver also contains a large number of immune cells called Kupffer cells. These cells act as a filter removing bacteria and other dangerous substances from the blood passing through the liver. Although we know and understand a great deal about how liver cells behave and function after transplant we have no idea what happens to the immune cells in the liver. These immune cells make up 85% of the total body reserves of these cells and serve an important function by clearing bacteria and bacterial products from the blood. A failure of these cells is associated with risk of infection. Infections, blood clotting disorders and many other serious medical issues are typical for patients suffering from chronic liver failure.

This study will use microscopic particles of a human protein called albumin in the form of microspheres to simulate bacteria in the blood. We can detect these microspheres by attaching a radioactive label to the spheres and measuring emission in a detector called a gamma counter. The level of radiation is quite small and similar to a bone scan. We have previously shown that healthy liver rapidly clears these albumin microspheres from the blood. We have also shown previously that after major liver surgery there is a delay in clearance of microspheres, which we believe equates to a poorly functioning innate immune system.

Liver transplantation is the only successful life-extending treatment for patients with chronic liver failure and cirrhosis. During liver transplantation it is known that a proportion of hepatocytes damaged and recover following the transplant. We want to establish the immediate particulate clearance capacity of the liver following transplantation and the pattern of recovery one week later. This is used as a surrogate for liver clearance of bacteria and bacterial products.

We also intend to measure the production of a set of proteins called acute phase proteins, which are produced by the liver and may be important in helping immune cells recognize bacteria. These proteins, also called opsonins, bind to the walls of bacteria and make it easier for immune cells to attach to the bacteria and eat them.

We also want to find out if there is any difference between non-marginal and marginal liver grafts and their reticuloendothelial clearance capacity. This study may provide important information regarding the need for post-operative antibiotics and prevention of infection in this patient group.

This research will be the first of its kind to address this issue in this vulnerable group of patients and no study has ever looked at the effect of transplantation on the immune cells of the liver. This study will investigate the ability of the liver to clear particles (albumin microspheres) from the blood and will monitor the recover and improvement in function of these cells over a period of time.

Results of any pilot studies

A study also from the eLISTER group (Edinburgh liver injury in surgery and transplantation experimental research) about the effect of major liver resection on innate immunity to bacterial endotoxin was approved by Lothian research Ethics Committee LREC/2002/1/31. This trial was performed between May 2003 and 2005. This study looked at the adaptive response of the reticuloendothelial system to major liver resection. We found a strong correlation between clearance of albumin microspheres and ICG (indocyanine green clearance), supporting the assertion that hepatocellular function and RES phagocytosis are related if only in terms of liver volume. We also demonstrated marked defects in RES phagocytosis in patients with chronic liver disease or normal liver function, who had undergone a major liver resection.

Validation of technique of measurement of phagocytic clearance of Tc-99m labelled (Nanocoll®) microaggregated human albumin To determine reticuloendothelial system (RES) phagocytosis activity and liver phagocytic function respectively we will measure plasma clearance of 99mTc labelled micro-aggregated human albumin without any imaging studies. It has been shown in several studies that this is a reliable method to estimate RES phagocytosis activity. By measuring the plasma radioactivity disappearance rate instead of doing imaging studies a radioactivity dose of less than 15 MBq is sufficient to determine 99mTc plasma clearance accurately. Disappearance of 99mTc blood activity will be measured serially at 3-minutes intervals to 30 minutes, at 10-minutes intervals to 60 minutes and at 20-minutes intervals to 120 minutes. Three half-life times required for the 99mTc albumin microspheres counting rate to fall from 100% to 50%, from 50% to 25% and from 25% to 12.5% of the value obtained at three minutes after injection are noted and the mean half-life and standard deviation, expressing the microspheres blood clearance, is calculated. To determine the possibly non-linear nature of albumin microspheres clearance over time the area under the curve will be calculated over the observation time using integral function. Mean half-life of albumin microspheres in the blood and area under the curve at day 1 and day 7 after transplantation will be expressed as a percentage of preoperative values and compared between individuals and patient groups. We hypothesize that the phagocytosis activity of marginal compared to good liver grafts is significantly impaired after liver transplantation due to the decreased number of phagocytes as well as due to the decreased synthesis of substances which usually facilitates phagocytosis. If this hypothesis is true, the RES phagocytosis activity in the marginal grafts should be significantly increased after liver transplantation and should be comparable to the RES phagocytosis activity of non-marginal grafts.

Aims

This project will test the hypothesis that liver transplantation of normal and marginal grafts results in a significant impairment of innate immunity to bacterial endotoxin.

We intend to characterise the nature or reticuloendothelial clearance impairment following liver transplantation and its recovery on marginal and non-marginal grafts. We also wish to correlate clearance capacity with measures of hepatocyte injury (ALT/AST) and liver dysfunction score to establish whether the two processes are independent or related.

In this regard we will compare marginal and non-marginal organs and the relationship between reticuloendothelial cell dysfunction and cold ischemic time. Reticuloendothelial clearance capacity will also be related to evidence of clinical infection in the postoperative course.

Research questions - Hypotheses

I. Liver transplantation results in a significant impairment of innate immunity to bacterial endotoxin.

II. The degree of impairment in innate immunity to endotoxin is directly related to the functional status of the liver graft. (Patients undergoing liver transplantation with non-marginal and marginal grafts will be compared).

III. To establish whether there is any correlation between liver cell (hepatocyte) injury and immune cell (Kupffer cell) injury after transplantation.

IV. To establish the effect of liver transplantation on serum expression of acute phase protein opsonins.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* chronic liver disease
* listed for transplantation at the Scottish Liver Transplant Unit

Exclusion Criteria:

* pregnancy (although pregnant patients would not be listed for liver transplant)
* prisoners
* acute liver failure
* living-related liver transplantation
* multi-organ transplantation or re-transplantation
* ABO incompatible donor
* HIV-positive donor or recipient
* not given informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on the waiting list for liver transplantation will be invited to participate in the study and written informed consent will be obtained from each participant. Patients who are undergoing transplantation will be studied before operation, 24 hours after transplantation and 7 days after transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
We want to establish the immediate particulate clearance capacity of the liver following transplantation and the pattern of recovery one week later. This is used as a surrogate for liver clearance of bacteria and bacterial products. | 7 days

SECONDARY OUTCOMES:
To establish whether there is any correlation between liver cell (hepatocyte) injury and immune cell (Kupffer cell) injury after transplantation. | 7 days
To establish the effect of liver transplantation on serum expression of acute phase protein opsonins. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Wigmore, Prof, MD, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, Midlothian, United Kingdom

REFERENCES:
- [Background] Schindl MJ, Millar AM, Redhead DN, Fearon KC, Ross JA, Dejong CH, Garden OJ, Wigmore SJ. The adaptive response of the reticuloendothelial system to major liver resection in humans. Ann Surg. 2006 Apr;243(4):507-14. doi: 10.1097/01.sla.0000205826.62911.a7. PMID 16552202
- [Background] Medzhitov R, Janeway C Jr. Innate immunity. N Engl J Med. 2000 Aug 3;343(5):338-44. doi: 10.1056/NEJM200008033430506. No abstract available. PMID 10922424